CLINICAL TRIAL: NCT05855876
Title: Reversal of Battle-Related Aging (ROBRA) in a Special Operations Forces Cohort
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Stella Center (Other)
Responsible Party: Principal Investigator, Eugene Lipov, Principal Investigator, Stella Center
Other Study IDs: ROBRA
Record Dates: First submitted 2023-04-21; First posted 2023-05-12 (Actual); Last update posted 2023-07-17 (Actual); Status verified 2023-07

CONDITIONS: Post-Traumatic Stress Disorder; Traumatic Brain Injury
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Brain Injuries, Traumatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Procedure: subanesthetic ketamine infusions and bilateral cervical sympathetic blocks — Combined protocol of subanesthetic ketamine infusions and bilateral cervical sympathetic blocks

SUMMARY:
The purpose of this study is to examine measures of GrimAge clock in SOF members undergoing treatment for PTSD/TBI using CSB.

DETAILED DESCRIPTION:
The primary objective of this study is to assess the impact of a combined protocol of subanesthetic ketamine infusions (SKI) and bilateral cervical sympathetic blocks (CSB) on aging, as measured by the GrimAge epigenetic clock.

The secondary objective of this study is to assess the impact of this treatment paradigm on PTSD and mental health, as measured over a 6 month time period using the following questionnaires: Post-traumatic Stress Disorder Checklist (PCL-5), Patient Health Questionnaire 9 (PHQ-9), Depressive Symptom Index-Suicidality Subscale (DSI-SS), Generalized Anxiety Disorder 7-item (GAD-7), and Neurobehavioral Symptom Inventory (NSI).

The tertiary objectives of the study are to investigate if PTSD is associated with significantly reduced free testosterone levels and increased C-reactive protein (CRP) levels.

ELIGIBILITY:
Inclusion Criteria:

* Recruited from SOF with an active duty history of at least 5 years.
* Subjects may be in active duty or retired, male and female, between the ages of 40 and 60 years old.
* The participants must have a confirmed diagnosis of PTSD, identified by Posttraumatic Stress Disorder Checklist for DSM-5 (PCL-5) scores higher than 40.
* The participants must have been on a stable pharmacological or psychotherapeutic therapy for at least three months (if applicable), and continue this treatment throughout the duration of the study.
* They must be able and willing to consent for the study. Individuals who are able to become pregnant must adhere to a medically accepted method of contraception (eg. hormonal birth control, barrier birth control, intrauterine device, abstinence).

Exclusion Criteria:

* Existing Horner syndrome;
* Allergy to local anesthetics or contrast;
* Previous history of stellate ganglion block with psychosis;
* Admission to in-patient psychiatric facility within last 3 months;
* History of moderate of severe TBI;
* Currently pregnant or breastfeeding;
* Current substance use disorder, or test positive for 1 or more illegal or controlled drugs on the initial urine drug screen, such as cocaine, marijuana, amphetamines, opioids, benzodiazepines, amongst others;
* Previous behavioral health diagnoses (bipolar I, psychosis, etc);
* Currently undergoing exposure therapy.

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: This study will include 20 individuals, recruited from SOF with an active duty history of at least 5 years. Subjects may be in active duty or retired, male and female, between the ages of 40 and 60 years old. The participants must have a confirmed diagnosis of PTSD.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2023-07-05 (Actual); Primary Completion 2024-04-05 (Estimated); Study Completion 2024-04-05 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in Epigenetic Aging at 15 days | day 15
  GrimAge epigenetic clock tool to assess DNA methylation
Change from baseline in Epigenetic Aging at 90 days | day 90
  GrimAge epigenetic clock tool to assess DNA methylation
Change from baseline in Epigenetic Aging at 180 days | day 180
  GrimAge epigenetic clock tool to assess DNA methylation

SECONDARY OUTCOMES:
Change from baseline in Post-Traumatic Stress Disorder (PTSD) symptoms at 15 days | day 15
  Post-traumatic Stress Disorder Checklist (PCL-5), a 20-item self-report measure yielding a total symptom severity score between 0 and 80.
Change from baseline in Post-Traumatic Stress Disorder (PTSD) symptoms at 90 days | day 90
  Post-traumatic Stress Disorder Checklist (PCL-5), a 20-item self-report measure yielding a total symptom severity score between 0 and 80.
Change from baseline in Post-Traumatic Stress Disorder (PTSD) symptoms at 180 days | day 180
  Post-traumatic Stress Disorder Checklist (PCL-5), a 20-item self-report measure yielding a total symptom severity score between 0 and 80.
Change from baseline in Depression at 15 days | day 15
  Patient Health Questionnaire 9 (PHQ-9), a 9-item self-report measure yielding a depression severity score between 0 and 27.
Change from baseline in Depression at 90 days | day 90
  Patient Health Questionnaire 9 (PHQ-9), a 9-item self-report measure yielding a depression severity score between 0 and 27.
Change from baseline in Depression at 180 days | day 180
  Patient Health Questionnaire 9 (PHQ-9), a 9-item self-report measure yielding a depression severity score between 0 and 27.
Change from baseline in Suicidal Ideation at 15 days | day 15
  Depressive Symptom Index-Suicidality Subscale (DSI-SS), a 4-item self-report measure yielding a suicidal ideation severity score between 0 and 12.
Change from baseline in Suicidal Ideation at 90 days | day 90
  Depressive Symptom Index-Suicidality Subscale (DSI-SS), a 4-item self-report measure yielding a suicidal ideation severity score between 0 and 12.
Change from baseline in Suicidal Ideation at 180 days | day 180
  Depressive Symptom Index-Suicidality Subscale (DSI-SS), a 4-item self-report measure yielding a suicidal ideation severity score between 0 and 12.
Change from baseline in Anxiety at 15 days | day 15
  Generalized Anxiety Disorder 7-item (GAD-7), a 7-item self-report measure yielding an anxiety severity score between 0 and 21.
Change from baseline in Anxiety at 90 days | day 90
  Generalized Anxiety Disorder 7-item (GAD-7), a 7-item self-report measure yielding an anxiety severity score between 0 and 21.
Change from baseline in Anxiety at 180 days | day 180
  Generalized Anxiety Disorder 7-item (GAD-7), a 7-item self-report measure yielding an anxiety severity score between 0 and 21.
Change from baseline in Post-Concussion Symptom Severity at 15 days | day 15
  Neurobehavioral Symptom Inventory (NSI), a 22-item self-report measure yielding a post-concussion symptom severity score between 0 and 88.
Change from baseline in Post-Concussion Symptom Severity at 90 days | day 90
  Neurobehavioral Symptom Inventory (NSI), a 22-item self-report measure yielding a post-concussion symptom severity score between 0 and 88.
Change from baseline in Post-Concussion Symptom Severity at 180 days | day 180
  Neurobehavioral Symptom Inventory (NSI), a 22-item self-report measure yielding a post-concussion symptom severity score between 0 and 88.
Change from baseline in Free testosterone levels at 15 days | day 15
  Quest diagnostics to measure Free testosterone levels
Change from baseline in Free testosterone levels at 90 days | day 90
  Quest diagnostics to measure Free testosterone levels
Change from baseline in Free testosterone levels at 180 days | day 180
  Quest diagnostics to measure Free testosterone levels
Change from baseline in C-reactive protein (CRP) levels at 15 days | day 15
  Quest diagnostics to measure C-reactive protein (CRP) levels
Change from baseline in C-reactive protein (CRP) levels at 90 days | day 90
  Quest diagnostics to measure C-reactive protein (CRP) levels
Change from baseline in C-reactive protein (CRP) levels at 180 days | day 180
  Quest diagnostics to measure C-reactive protein (CRP) levels

CONTACTS AND LOCATIONS:
Overall Officials: Eugene Lipov, MD, Principal Investigator — Stella Center
Locations (1):
- Stella Center, Westmont, Illinois, United States